CLINICAL TRIAL: NCT07226713
Title: A Single-Arm, Open-label, Phase II Study Evaluating Pacritinib in Participants With Metastatic Castrate-Resistant Prostate Cancer That Progressed on or After Prior Treatment With Androgen Receptor Signaling Inhibitors - (POSTPONE)
Brief Title: Pacritinib in Participants With Metastatic Castrate-Resistant Prostate Cancer That Progressed on or After Prior Treatment With Androgen Receptor Signaling Inhibitors
Acronym: POSTPONE
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Medical College of Wisconsin (Other)
Responsible Party: Principal Investigator, Deepak Kilari, Associate Professor, Medical College of Wisconsin
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIT-KILARI-POSTPONE
Record Dates: First submitted 2025-11-06; First posted 2025-11-10 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-11

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — 11-(2-pyrrolidin-1-ylethoxy)-14,19-dioxa-5,7,26-triazatetracyclo(19.3.1.1(2,6).1(8,12))heptacosa-1(25),2(26),3,5,8,10,12(27),16,21,23-decaene

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Pacritinib (Experimental): Pacritinib is an oral drug.
  Interventions: Drug: Pacritinib

INTERVENTIONS:
Drug: Pacritinib — Pacritinib is an oral drug which will be taken daily at a dose of 200 mg twice a day (BID).
  Other Names: SB1518

SUMMARY:
This is a single-arm, open-label phase 2 study to evaluate the role of pacritinib for patients with metastatic castrate-resistant prostate cancer that have progressed on ARSI. Patients will receive pacritinib 200 mg twice daily. To be eligible, patients must have a biopsy of a metastatic site within 30 days of treatment that demonstrates positive STAT5 activation status

ELIGIBILITY:
Inclusion Criteria:

I. To be eligible for screening:

1. Patients aged ≥ 18 years.
2. Histologically or cytologically confirmed prostate adenocarcinoma.
3. Have current evidence of metastatic disease documented by either bone scan, CT/MRI and/or PSMA PET scan
4. Have disease that progressed while receiving androgen deprivation therapy (ADT) (or post bilateral orchiectomy) and during or after treatment with at least one androgen receptor signaling inhibitor (ARSI) (e.g., abiraterone acetate, enzalutamide, apalutamide, darolutamide) for metastatic hormone-sensitive prostate cancer (HSPC) (mHSPC or nmHSPC) or mCRPC.

   a. Note: Participants may have received abiraterone acetate and docetaxel or darolutamide and docetaxel for HSPC. However, participants must have received no more than 6 cycles of docetaxel and had no radiographic disease progression while receiving docetaxel. Disease progression could be prostate-specific antigen (PSA) based or radiographic progression per Prostate Cancer Working Group 3 (PCWG3) guidelines.
5. Screening serum testosterone < 50 ng/dL.
6. Eastern Cooperative Oncology Group (ECOG), Performance Status grade 0-1 or Karnofsky Performance Status ≥ 70
7. No prior janus kinase2 (JAK2) inhibitor treatment.
8. Left ventricular cardiac ejection fraction of ≥ 50% by echocardiogram or multigated acquisition (MUGA) scan.
9. Adequate organ function as defined by the following laboratory values at screening:

   1. Serum aspartate transaminase (AST), serum glutamic oxaloacetic transaminase (SGOT), serum alanine transaminase (ALT) and serum glutamic pyruvic transaminase (SGPT) < 2.5 x upper limit of normal (ULN).
   2. Total serum bilirubin ≤ 1.5 x ULN. In subjects with Gilbert's syndrome, if total bilirubin is >1.5 × ULN, measure direct and indirect bilirubin and if direct bilirubin is ≤ 1.5 × ULN, the subject may be eligible).
   3. Serum potassium ≥ 3.5 mmol/L. Supplementation and re-screening is allowed.
   4. Estimated glomerular filtration rate (GFR) > 45 ml/min using the Cockroft-Gault equation.
   5. Platelets ≥ 100,000/mL independent of transfusion and/or growth factors within three months
   6. Hemoglobin ≥ 9.0 g/dL independent of transfusion and/or growth factors within three months
   7. Absolute neutrophil count ≥ 500/µL.
   8. Serum albumin ≥ 3.0 g/dL.
   9. Adequate coagulation defined by prothrombin time (PT)/international normalized ratio (INR) and PTT ≤ 1.5 ULN.
10. Male patients, even if surgically sterilized (i.e., status post-vasectomy), must agree to one of the following:

    a. Practice effective barrier contraception and another effective method of birth control if he is having sex with a woman of childbearing potential during the entire study period and through 30 calendar days after the last dose of study agent
11. Ability to understand a written informed consent document, and the willingness to sign it.

II. To be eligible for treatment:

1. Patients must meet all screening criteria described above.
2. Patients must provide tumor tissue from a fresh core or excisional biopsy from soft tissue not previously irradiated. Samples from tumors progressing at a prior site of radiation are allowed. Participants with bone-only or bone-predominant disease may provide a bone biopsy sample. A tumor sample must be obtained within 30 days of treatment.
3. STAT5 activation levels need to be high, with positive STATA5 activation status defined as detectable nuclear localized Stat5 in >5% of cancer cells from tissue obtained within 30 days of treatment.

Exclusion Criteria:

1. Patient does not have positive STAT5 activation status in PC core biopsies.
2. Previously treated with pacritinib.
3. Use of investigational agents within 28 days prior to randomization.
4. Use of other prohibited medications within seven days prior to Cycle 1, Day 1 or 5x half-life of the drug, whichever is longer.
5. Systemic treatment with a strong CYP3A4 inhibitor or inducer within 14 days prior to the start of treatment.
6. Uncontrolled hypertension.
7. Baseline severe hepatic impairment (Child-Pugh Class B & C).
8. An intercurrent illness that is not controlled, such as active infection, psychiatric illness, or social situations that would limit compliance with study requirements.
9. Any chronic medical condition requiring a higher dose of corticosteroid than an equivalent of 10 mg prednisone/prednisolone per day.
10. Significant recent bleeding history, as defined as National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) v5.0 Grade ≥ 2 within three months prior to start of treatment, unless precipitated by an inciting event (e.g., surgery, trauma, or injury).
11. Systemic treatment with medications that increase the risk of bleeding, including anticoagulants (warfarin, direct oral anticoagulant, etc.), antiplatelet agents (except for aspirin dosages of ≤ 100 mg/day), anti-vascular endothelial growth factor (anti-VEGF) agents, and daily use of COX-1 inhibiting nonsteroidal anti-inflammatory agents (NSAIDs) within 14 days prior to the start of treatment.
12. Systemic treatment with medications that can prolong the QT interval within 14 days prior to the start of treatment. Shorter washout periods may be permitted with the approval of the PI, provided that the washout period is at least five half-lives of the drug prior to the start of treatment.
13. Any history of CTCAE v5.0 Grade ≥ 2 cardiac conditions within six months before treatment Day 1. Patients with asymptomatic Grade 2 non-dysrhythmia cardiovascular conditions may be considered for inclusion, with the approval of the principal investigator, if stable and unlikely to affect patient safety.
14. QT corrected for heart rate by Fridericia's cube root formula (QTcF) prolongation > 450 ms or other factors that increase the risk for QT interval prolongation (e.g., heart failure, hypokalemia [defined as serum potassium < 3.0 mEq/L that is persistent and refractory to correction]), or history of long QT interval syndrome.
15. New York Heart Association Class II, III, or IV congestive heart failure.
16. Any active gastrointestinal or metabolic condition that could interfere with absorption of oral medication.
17. Active or uncontrolled inflammatory or chronic functional bowel disorder, such as Crohn's disease, inflammatory bowel disease, chronic diarrhea, or chronic constipation.
18. Other malignancy within three years prior to the start of treatment, other than curatively treated basal cell or squamous cell skin
19. Uncontrolled intercurrent illness, including, but not limited to, ongoing active infection, psychiatric illness, or social situation that, in the judgment of the treating physician, would limit compliance with study requirements.
20. Known seropositivity for human immunodeficiency virus.
21. Known active hepatitis A, B, or C virus infection.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2029-03-01 (Estimated); Study Completion 2031-03-01 (Estimated)

PRIMARY OUTCOMES:
Progression-free Survival | Six months
  Six-month radiographic progression-free survival is defined as the probability that a given subject will be alive and free from radiographic progression per Prostate Cancer Working Group 3 guidelines at 24 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Deepak Kilari, MD, Principal Investigator — Medical College of Wisconsin
Locations (1):
- Froedtert & the Medical College of Wisconsin, Milwaukee, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No